CLINICAL TRIAL: NCT04449172
Title: ProtocoL for GFR Measurement Using Iohexol (SCOPE-PLUS) - A Substudy of the SCOPE Study
Acronym: SCOPE-PLUS
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Erasmus Medical Center (Other); Institut Catala de Salut (Other Government); Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_05_2019; Grant Agreement n. 634869 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2020-06

CONDITIONS: Chronic Kidney Diseases
Keywords: glomerular filtration rate; older people; ioexol
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SCOPE-PLUS is an optional substudy of the observational SCOPE Study (Screening for Chronic Kidney Disease among Older People across Europe, NCT02691546). The objective of the SCOPE-PLUS study is to derive new equations based on innovative and novel biomarkers of CKD function and compare its accuracy to measure GFR in the population older than 75 years.

DETAILED DESCRIPTION:
SCOPE-PLUS is an optional substudy of the SCOPE cohort study (Screening for Chronic Kidney Disease among Older People across Europe, NCT02691546). SCOPE has retrieved data on a wide panel of biomarkers of CKD in a large study cohort enrolling about 2,450 older people in Italy, Spain, Germany, Austria, Netherlands, Poland and Israel. The innovative biomarkers have been already validated by the literature, and include e.g. Cystatin C (CysC), β-Trace protein (BTP), and Beta2-microglobulin. Others promising novel biomarkers of CKD, based on metabolomic and proteomic determinations or other techniques have been evaluated. The objective of the SCOPE-plus study is to to verify the accuracy of newly developed equations based on innovative and novel biomarkers of CKD function by calculating the percentage of estimates within 30% (P30) of the measured GFR (mGFR). The mGFR will be obtained by the assessment of nonradioactive iohexol clearance. Patients previously enrolled in the SCOPE study, are invited to participate in this additional protocol. Iohexol is an iodinated contrast medium with characteristics similar to those of inulin, being freely filtered by the glomerulus, neither secreted nor reabsorbed by the renal tubules and recovered almost 100% in the urine. These characteristics made it an ideal agent for the determination of the renal function.

ELIGIBILITY:
Inclusion Criteria:

* to be eligible for this study, subjects must have been enrolled in the SCOPE study

Exclusion Criteria for substudy:

* a thyroid-stimulating hormone level less than 0.3 mlU/L
* a known iodine allergy
* oedema
* ascites
* clinically symptomatic heart failure

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: subjects with 75 years or older previously enrolled in the SCOPE study (NCT02691546)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
To measure GFR in subjects aged 75 or older by iohexol clearance to verify the accuracy of equations of innovative and novel biomarkers of CKD newly evaluated in the SCOPE study | 300 minutes from intravenous injection of iohexol
  Iohexol solution 5 mL (Omnipaque, GE Healthcare), containing 3235 mg of iohexol will be administered intravenously into an antecubital, forearm, or hand vein and flushed with 10 mL of normal saline. Blood samples for serum creatinine and other biomarkers will be obtained before iohexol is applied. Blood samples will be obtained after 5 minutes from the contralateral arm to confirm that the Iohexol has been administered correctly intravenously. Subsequent blood sample will be collected (always from the contralateral arm) at 10, 20, 30, 45, 60, 90, 120, 180, 240 and 300 minutes after injection. The exact timing of the samples collection will be recorded. All clearance measurements will be started between 8:00 and 10:30 a.m.

CONTACTS AND LOCATIONS:
Locations (5):
- MEDIZINISCHE UNIVERSITAT- Internal Medicine/Nephrology/Geriatric Department, Graz, Austria
- Italy (2):
  - INRCA Research Hospital, Ancona
  - INRCA Research Hospital, Cosenza
- ERASMUS UNIVERSITAIR MEDISCH CENTRUM-Department of Internal Medicine, Rotterdam, Netherlands
- INSTITUT CATALA DE LA SALUT-Internal Medicine Deparment, Barcelona, Spain